CLINICAL TRIAL: NCT00148915
Title: A One Year, Parallel, Placebo-controlled, Double-blind, Randomized Study to Assess the Effect of Monthly 150 mg Oral Ibandronate Dosing Versus Placebo on Bone Quality and Strength at the Proximal Femur in Women With Osteoporosis
Brief Title: A Study To Assess the Quality and Strength of Bone in Women Participants With Osteoporosis Taking Oral Ibandronate Versus Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BON103593
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; bisphosphonates; bone
MeSH Terms: conditions — Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibandronate (Experimental): Participants will receive 150 milligrams (mg) ibandronate tablet orally once monthly for one year.
  Interventions: Drug: ibandronate
- Placebo (Placebo Comparator): Participants will receive ibandronate matched placebo tablet orally once monthly for one year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ibandronate
  Other Names: Boniva
  Arms: Ibandronate
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study is to estimate the effect of oral ibandronate sodium (Boniva) taken once monthly versus placebo on bone quality and strength at the proximal femur at one year.

ELIGIBILITY:
Inclusion criteria:

* Ambulatory, postmenopausal women between the age of 55 to 80 years diagnosed with osteoporosis
* BMD T-Score less than or equal to (<=) -2.0 at total spine or total femur or total neck, and BMD T-score greater than or equal to (>=) -5.0 at all 3 sites

Exclusion criteria:

* Have been treated with other bisphosphonates or using chronic steroids within the past 6 months
* Have a history of major upper gastrointestinal (GI) diseases or have severe kidney dysfunction
* Have a spine fracture (identified on X-ray)

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Mean percent change in integral (cortical and trabecular bone compartments combined) hip bone mineral density (BMD) as determined by Volumetric Quantitative Computed Tomography (vQCT) at one year | Year 1

SECONDARY OUTCOMES:
Mean percent change in BMD of the proximal femur and lumbar spine according to vQCT at one year | Year 1
Mean percent change of proximal femur and spine BMD according to Dual- Energy X-ray Absorptiometry (DXA) scans | Year 1
Hip geometry assessed by cross-sectional dimensions of hip using vQCT | Year 1
Finite element composition of hip and spine to estimate hip and spine strength | Year 1
Hip geometry assessed by cross-sectional dimensions of hip using DXA | Year 1
Trabecular bone dimensions by bone biopsies using histomorphometry and micro computed tomography to assess bone quality | Year 1
Change from baseline for serum-C-terminal cross-linking telopeptide of Type I collagen (Serum-CTX) | Months 3, 6, 9, and 12
Change from baseline for bone-specific alkaline phosphatase (Bone ALP) | Months 3, 6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: HoffmannLaRoche Clinical Trials, MD, Study Director — Hoffmann-La Roche
Locations (13):
- United States (13):
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Bathesda, Maryland
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, West Haverstraw, New York
  - GSK Investigational Site, Duncansville, Pennsylvania